CLINICAL TRIAL: NCT06241651
Title: Conduction System Pacing Versus Biventricular Pacing for Heart Failure Patients with Right Ventricular Pacing Upgraded to Cardiac Resynchronization Therapy: a Prospective Multicenter Non-inferiority Randomized Controlled Study
Brief Title: CSP Versus BiVP for Heart Failure Patients with RVP Upgraded to Cardiac Resynchronization Therapy
Acronym: CSP-UPGRADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Soochow University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Third Affiliated Hospital of Soochow University (Other); Rugao People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shantou Central Hospital (Other); Meizhou People's Hospital (Other); Changzhou Second People's Hospital affiliated with Nanjing Medical University (Other); Zhangjiagang First People's Hospital (Other); Huizhou Third People's Hospital, Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jiangang Zou, Head of Internal Medicine, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-811
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Conduction System Pacing; Biventricular Pacing; Cardiac Resynchronization Therapy; Right Ventricular Pacing; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CSP group (Experimental): In this group, CSP lead is attempted to be placed, including LBBP and HBP.
  Interventions: Device: Conduction system pacing
- BiVP group (Active Comparator): In this group, traditional RA lead , RV lead and LV lead are attempted to be placed.
  Interventions: Device: Biventricular pacing

INTERVENTIONS:
Device: Conduction system pacing — Firstly, we will attempt LBBP if the patient is allocated to the experimental group. If we can not achieve LBBP successfully, then we will turn to attempt HBP.
  Arms: CSP group
Device: Biventricular pacing — Implantation of RA lead, RV lead and LV lead are attempted using the standard-of-care technique.
  Arms: BiVP group

SUMMARY:
The present study is a prospective, multicenter, non-inferiority, randomized controlled trail. It aims to investigate whether the efficacy of conduction system pacing (CSP) is non-inferior to biventricular pacing (BiVP) in patients with heart failure and right ventricular pacing (RVP) requiring upgrading to cardiac resynchronization therapy (CRT).

DETAILED DESCRIPTION:
RVP is a standardized treatment strategy for severe bradyarrhythmia. However, RVP can result in electrical and mechanical dyssynchrony of the heart, which will adversely affect cardiac function. Until now, many studies have shown that RVP can promote the progression of heart failure, especially in patients with high ventricular pacing percentage. For these heart failure patients, upgrading to CRT is a feasible and effective therapy.

BiVP is a traditional method to achieve CRT, which can improve cardiac synchrony and provide great clinical outcomes for heart failure patients upgraded from RVP. CSP contains left bundle branch pacing (LBBP) and His bundle pacing (HBP), which is able to activate native His-Purkinje conduction system and solve the problems caused by RVP. Although HBP has high technical requirements, lower sense value and higher threshold, it is the pacing modality closest to physiological conditions so far. Since first reported by Huang et al. in 2017, LBBP has been carried out boomingly all over the world. LBBP has been reported to offer higher success rate with higher sense value and lower pacing thresholds compared with HBP, which can also achieve similar electrical and mechanical resynchronization as well as HBP.

However, no randomized controlled studies have been reported to compare the efficacy of CSP and BiVP in patients with heart failure and RVP requiring upgrading to CRT. CSP-UPGRADE is a non-inferiority study, and the purpose of which is to investigate whether the efficacy of CSP is not inferior to BiVP in such patients. Eligible patients will be 1:1 randomized to two groups. The primary outcome is change in LVEF between baseline and six months after device implantation assessed by echocardiography. According to BUDAPEST-CRT Upgrade trial, half of lower limit of the 95% confidence interval for difference in mean ΔLVEF between the CRTD and ICD group is about 3.8%, which is used as non-inferiority margin in the present study. Based on previous studies and cases, it is assumed that the mean ΔLVEF values in patients upgraded to CSP and BiVP are equal and the standard deviations are both 5%. With power as 80%, alpha as 0.025, rate of lost-of-follow-up as 10%, the final sample size was estimated as 66 by using PASS Version 21.0.3 (33 patients for each group). If the non-inferiority test reaches positive results, then we will further verify whether CSP is superior to BiVP in such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic heart failure (LVEF <50%) after right ventricular pacing for at least 3 months;
2. NYHA class II-IV;
3. NT-proBNP >125pg/mL in patients with sinus rhythm, NT-proBNP >250pg/mL in patients with atrial fibrillation;
4. Right ventricular pacing percentage >40%;
5. Adult patients aged 18-80;
6. With informed consent signed.

Exclusion Criteria:

1. History of acute myocardial infarction within 3 months before enrollment;
2. Frequent premature ventricular contraction (>15%) or malignant ventricular arrhythmia which is difficult to control;
3. History of valvular heart disease intervention within 3 months before enrollment;
4. After mechanical tricuspid valve replacement;
5. Ventricular septal hypertrophy (≥15mm during diastole);
6. Complex congenital heart disease;
7. History of heart transplantation;
8. Enrollment in any other study;
9. Pregnant or with child-bearing plan;
10. A life expectancy of less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
ΔLVEF | Baseline; 6-month follow-up
  Change in LVEF between baseline and six months after device implantation

SECONDARY OUTCOMES:
ΔLVEDD | Baseline; 3-month follow-up; 6-month follow-up
  Change in LVEDD between baseline and follow-up
ΔLVEDV | Baseline; 3-month follow-up; 6-month follow-up
  Change in LVEDV between baseline and follow-up
ΔLVESV | Baseline; 3-month follow-up; 6-month follow-up
  Change in LVESV between baseline and follow-up
Paced QRS duration | 1 day before discharge; 1-month follow-up; 3-month follow-up; 6-month follow-up
  Paced QRS duration is evaluated before discharge and follow-up
Echocardiographic response rate | Baseline; 6-month follow-up
  The percentage of patients responding to CRT upgrade assessed by echocardiography
Changes in NT-proBNP | Baseline; 3-month follow-up; 6-month follow-up
  The changes of NT-proBNP between baseline and follow-up
Changes in New York Heart Association Heart Function Classification | Baseline; 1-month follow-up; 3-month follow-up; 6-month follow-up
  The higher the classification, the more severe the heart failure symptoms (four levels: I, II, III and IV)
Changes in 6-minute Walk Distance | Baseline; 3-month, 6-month follow-up
  Distance that a participant walk within 6 minutes
Change in Quality Of Life Questionnaire score | Baseline; 3-month follow-up; 6-month follow-up
  Reflect the effect of heart failure on quality of life, and higher scores represent a worse outcome
Incidence of clinical adverse events | 1 day before discharge; 1-month follow-up; 3-month follow-up; 6-month follow-up
  Including all-cause mortality, cardiovascular mortality, heart failure hospitalization and malignant ventricular arrhythmia
Procedure-related costs | 1 day before discharge
  Costs related to device implantation
Estimated longevity of the device | 1 day before discharge; 1-month follow-up; 3-month follow-up; 6-month follow-up
  The longevity of the device will be estimated during pacemaker test
Pacing parameters | 1 day before discharge; 1-month follow-up; 3-month follow-up; 6-month follow-up
  Number of atrial fibrillation and NSVT/VT
Pacemaker related complications | 1 day before discharge; 1-month follow-up; 3-month follow-up; 6-month follow-up
  Including but not limited to hemorrhage, pneumothorax, pericardial effusion, device-related infection and lead displacement

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Chung MK, Patton KK, Lau CP, Dal Forno ARJ, Al-Khatib SM, Arora V, Birgersdotter-Green UM, Cha YM, Chung EH, Cronin EM, Curtis AB, Cygankiewicz I, Dandamudi G, Dubin AM, Ensch DP, Glotzer TV, Gold MR, Goldberger ZD, Gopinathannair R, Gorodeski EZ, Gutierrez A, Guzman JC, Huang W, Imrey PB, Indik JH, Karim S, Karpawich PP, Khaykin Y, Kiehl EL, Kron J, Kutyifa V, Link MS, Marine JE, Mullens W, Park SJ, Parkash R, Patete MF, Pathak RK, Perona CA, Rickard J, Schoenfeld MH, Seow SC, Shen WK, Shoda M, Singh JP, Slotwiner DJ, Sridhar ARM, Srivatsa UN, Stecker EC, Tanawuttiwat T, Tang WHW, Tapias CA, Tracy CM, Upadhyay GA, Varma N, Vernooy K, Vijayaraman P, Worsnick SA, Zareba W, Zeitler EP. 2023 HRS/APHRS/LAHRS guideline on cardiac physiologic pacing for the avoidance and mitigation of heart failure. Heart Rhythm. 2023 Sep;20(9):e17-e91. doi: 10.1016/j.hrthm.2023.03.1538. Epub 2023 May 20. PMID 37283271
- [Background] Tops LF, Schalij MJ, Bax JJ. The effects of right ventricular apical pacing on ventricular function and dyssynchrony implications for therapy. J Am Coll Cardiol. 2009 Aug 25;54(9):764-76. doi: 10.1016/j.jacc.2009.06.006. PMID 19695453
- [Background] Kaye GC, Linker NJ, Marwick TH, Pollock L, Graham L, Pouliot E, Poloniecki J, Gammage M; Protect-Pace trial investigators. Effect of right ventricular pacing lead site on left ventricular function in patients with high-grade atrioventricular block: results of the Protect-Pace study. Eur Heart J. 2015 Apr 7;36(14):856-62. doi: 10.1093/eurheartj/ehu304. Epub 2014 Sep 4. PMID 25189602
- [Background] Khurshid S, Obeng-Gyimah E, Supple GE, Schaller R, Lin D, Owens AT, Epstein AE, Dixit S, Marchlinski FE, Frankel DS. Reversal of Pacing-Induced Cardiomyopathy Following Cardiac Resynchronization Therapy. JACC Clin Electrophysiol. 2018 Feb;4(2):168-177. doi: 10.1016/j.jacep.2017.10.002. Epub 2017 Nov 15. PMID 29749933
- [Background] Shan P, Su L, Zhou X, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA, Huang W. Beneficial effects of upgrading to His bundle pacing in chronically paced patients with left ventricular ejection fraction <50. Heart Rhythm. 2018 Mar;15(3):405-412. doi: 10.1016/j.hrthm.2017.10.031. Epub 2017 Nov 16. PMID 29081396
- [Background] Qian Z, Wang Y, Hou X, Qiu Y, Wu H, Zhou W, Zou J. Efficacy of upgrading to left bundle branch pacing in patients with heart failure after right ventricular pacing. Pacing Clin Electrophysiol. 2021 Mar;44(3):472-480. doi: 10.1111/pace.14147. Epub 2021 Jan 31. PMID 33372293
- [Background] Merkely B, Hatala R, Wranicz JK, Duray G, Foldesi C, Som Z, Nemeth M, Goscinska-Bis K, Geller L, Zima E, Osztheimer I, Molnar L, Karady J, Hindricks G, Goldenberg I, Klein H, Szigeti M, Solomon SD, Kutyifa V, Kovacs A, Kosztin A. Upgrade of right ventricular pacing to cardiac resynchronization therapy in heart failure: a randomized trial. Eur Heart J. 2023 Oct 21;44(40):4259-4269. doi: 10.1093/eurheartj/ehad591. PMID 37632437